CLINICAL TRIAL: NCT03562221
Title: Prevention of Celiac Disease in Skåne (in Swedish - Prevention av Celiaki i Skåne)
Brief Title: Prevention of Celiac Disease in Skåne
Acronym: PreCiSe
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lund University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2018/61
Record Dates: First submitted 2018-05-21; First posted 2018-06-19 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Celiac Disease in Children
Keywords: coeliac disease; celiac disease autoimmunity
MeSH Terms: conditions — Celiac Disease | interventions — Diet, Gluten-Free; Probiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Gluten free diet (Experimental): Gluten free diet
  Interventions: Other: Gluten free diet
- Probiotics (Active Comparator): Capsules with a combination of two probiotic bacteria with maize starch as excipient and at a total dose of 10(10) colony forming units (CFU)/capsule.
  Interventions: Dietary Supplement: Probiotics
- Placebo (Placebo Comparator): Placebo capsules with maize starch and without any bacteria.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Other: Gluten free diet — Controlled gluten free diet
  Arms: Gluten free diet
Dietary Supplement: Probiotics — Capsules
  Arms: Probiotics
Dietary Supplement: Placebo — Capsules
  Arms: Placebo

SUMMARY:
This study aims to investigate the impact of being on a gluten free diet the first three years of life compared to a daily intake of a probiotic supplementation or placebo on the risk of developing celiac disease autoimmunity or celiac disease in genetically susceptible children.

This is a three-arm (1:1:1) randomized trial where study participants are randomly allocated to one of the three study groups before the age of 4 months. Regular clinical visits (4 times/year) during the intervention phase and yearly there after, up to the age of 7 years.

DETAILED DESCRIPTION:
The primary hypothesis to be tested is that a strictly gluten free diet during the first three years of life with a slow introduction of gluten during the follow-up period will induce tolerance to gluten. A similar hypothesis is tested if a daily supply of two different lactobacillus (LB) strains can suppress an inflammatory response to gluten in the intestine by stimulating regulatory T-cells and reduced permeability of gluten peptides in the intestine.

The secondary hypothesis tested is that celiac disease can not be prevented, but the onset of the disease will be delayed in children returning to a gluten-containing diet after the intervention period (gluten free diet) or probiotic treatment) during the first three years of life. The intervention period is 3 years and the follow-up period is further 4 years.

The primary aim is to study the proportion of children who develop celiac disease autoimmunity and progression to celiac disease by the age of 3 years. Secondary aim is to study the proportion of children who developed celiac disease at the age of 7 years.

ELIGIBILITY:
Inclusion Criteria:

* Children screened positive for human leucocyte antigen (HLA) DR3-DQ2/DR3-DQ2
* Children must be enrolled to the study by 4 months of age (before gluten consumption has started).

Exclusion Criteria:

* Congenital chronic disorder where intervention with diet or probiotics may be affected.
* Written consent from both caregivers are missing

Ages: 4 Months to 4 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 220 (Actual)
Dates: Start 2018-12-04 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Number of children tested positive for persistent tissue transglutaminase (tTG) autoantibodies, defined as celiac disease autoimmunity | from 4 months of age up until 7 years of age
  Radioligand binding assays (RBA) will be used to measure tTG autoantibodies in serum samples collected every third months up until the age of 3 years and then annually up until the age of 7 years.

SECONDARY OUTCOMES:
Number of children diagnosed with celiac disease | Up until 7 years of age
  A celiac disease diagnose will be defined by an intestinal biopsy showing a Marsh score of 2 or higher or by high levels of tTG autoantibodies (> 100 units) in at least 2 consecutive blood samples.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Agardh, PhD, Principal Investigator — Lund University
Locations (1):
- Clinical Research Center (CRC), Bldng 60:11, Malmo, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Af Segerstad EMH, Ericson-Hallstrom E, Bokstrom A, Armeni M, Savolainen O, Andren Aronsson C. Plasma Alkylresorcinols Is an Objective Biomarker for Gluten Intake in Young Children. J Nutr. 2025 Mar;155(3):985-993. doi: 10.1016/j.tjnut.2025.01.020. Epub 2025 Jan 27. PMID 39880171